CLINICAL TRIAL: NCT04963140
Title: Optimal Self-Management Of Asthma By Forced Oscillation Technique: a Randomised Controlled Trial
Brief Title: Self-Management Of Asthma By Forced Oscillation Technique
Acronym: PIANOFORTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Restech Srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1/20
Record Dates: First submitted 2021-06-18; First posted 2021-07-15 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2022-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention subjects will monitor their lung function daily by Forced Oscillation Technique (FOT) device. The embedded algorithm signals when an increased risk of exacerbation is detected and subjects shall modify their treatment based on the action plan prescribed by the study doctor at enrolment and used for the self-management of their asthma
  Interventions: Other: Optimized self-management of asthma
- Control (Sham Comparator): Control subjects will monitor their lung function daily by Forced Oscillation Technique (FOT) device. The embedded algorithm used in the intervention arm is disabled. Subjects will follow the action plan prescribed by the study doctor at enrolment for the self-management of their asthma
  Interventions: Other: Conventional self-management of asthma

INTERVENTIONS:
Other: Optimized self-management of asthma — Short-term increase of asthma medication (as prescribed by the study doctor at enrolment) if an increased risk of asthma exacerbations is detected by the home monitoring device
  Arms: Intervention
Other: Conventional self-management of asthma — Short-term increase of asthma medication (as prescribed by the study doctor at enrolment) is based on subject's self-perception of symptoms
  Arms: Control

SUMMARY:
Self-management strategies for asthma, including patients engagement and adherence to personalised action plans with advice on recognizing and responding to deterioration in control with effective treatments can improve asthma outcomes and possibly reduce the risk of future exacerbations. However, the real-life evidence is that asthma control remains sub-optimal in the majority of cases, thus increasing the related socio-economic costs worldwide.

Because an increased variability of lung function remains a hallmark of poor asthma control and exacerbations, its assessment over time could contribute to the success of self-management plans. Previous studies have shown the potential of Forced Oscillation Technique (FOT) as a tool for monitoring increased variability of airway obstruction and for identifying the onset of acute deterioration of airway function.

The aim of this study is to test the hypothesis that a personalised self-management plan including FOT improves asthma control and reduces number of days with increased symptoms compared to conventional asthma treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6-65 years old
* Diagnosis of persistent asthma
* Treatment level at study entry:

  * For children 6-11 years: Step2 or Step3 of the GINA document
  * For adolescents and adults 12-65 years: Step2 under daily low-dose inhaled corticosteroids (ICS), Step 3 or Step 4 of the GINA document
* Uncontrolled asthma (ACQ-5 > 1.5) that, according to the physician, does not warrant an immediate step-up of the treatment
* History of moderate or severe exacerbations in the twelve (12) months prior to baseline visit

Exclusion Criteria:

* Use of oral, rectal or parenteral glucocorticosteroids 30 days before enrolment
* Treatment with leukotriene receptor antagonist (LTRA)
* Treatment with maintenance and reliever therapy (SMART/MART)
* Smoking, current or previous with a history of 10 pack-years or more
* Documented COPD or other concomitant clinically important diseases or cognitive impairment that, according to the physician, may interfere with the subject's ability or safety to participate in the study
* Obesity (for subjects 6-19 years: BMI ≥ 95th percentile; for adults 20-65 years: BMI ≥ 40kg⋅m-2
* For school-age children (6-11 years old): gestational age at birth < 37 weeks or documented bronchopulmonary dysplasia (BPD)
* Prolonged absence from home during the monitoring period (i.e. at recruitment, expected ≥3 consecutive weeks for ≥2 times during the 9- month monitoring period) Subject currently enrolled in other clinical trials related or involving the study of the respiratory system
* History of near-fatal asthma
* Women who are pregnant, nursing or intending to become pregnant during the time of the study
* Absence of health insurance coverage (applies to French centres only)

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Asthma Control | 6 months from enrolment
  Change of percentage of subjects who improve their Asthma Control Questionnaire (ACQ-5)
Symptoms | From month no. 2 through study completion, an average of 7 months
  Change of percentage of days with non-increased symptoms from baseline

SECONDARY OUTCOMES:
Asthma Control | 3 months from enrolment
  Change of percentage of subjects who improve their Asthma Control Questionnaire (ACQ-5)
Asthma Control | 9 months from enrolment
  Change of percentage of subjects who improve their Asthma Control Questionnaire (ACQ-5)
Asthma Control | 3 months from enrolment
  Change of percentage of subjects who improve their Asthma Control Questionnaire (ACQ-5) moving from uncontrolled to controlled asthma
Asthma Control | 6 months from enrolment
  Change of percentage of subjects who improve their Asthma Control Questionnaire (ACQ-5) moving from uncontrolled to controlled asthma
Asthma Control | 9 months from enrolment
  Change of percentage of subjects who improve their Asthma Control Questionnaire (ACQ-5) moving from uncontrolled to controlled asthma
Asthma Control | 3 months from enrolment
  Change of percentage of adolescent and adult subjects (12+ years old) who improve their Asthma Control Questionnaire (ACQ-5)
Asthma Control | 6 months from enrolment
  Change of percentage of adolescent and adult subjects (12+ years old) who improve their Asthma Control Questionnaire (ACQ-5)
Asthma Control | 9 months from enrolment
  Change of percentage of adolescent and adult subjects (12+ years old) who improve their Asthma Control Questionnaire (ACQ-5)
Asthma Control | 3 months from enrolment
  Change of mean Asthma Control Questionnaire (ACQ-5); the expected ACQ-5 range is 0 - 3.5, with lower values indicating better asthma outcome
Asthma Control | 6 months from enrolment
  Change of mean Asthma Control Questionnaire (ACQ-5); the expected ACQ-5 range is 0 - 3.5, with lower values indicating better asthma outcome
Asthma Control | 9 months from enrolment
  Change of mean Asthma Control Questionnaire (ACQ-5); the expected ACQ-5 range is 0 - 3.5, with lower values indicating better asthma outcome
Exacerbation | Through study completion, an average of 9 months
  Change of number of moderate and severe exacerbations
Controller medication usage | From month no. 2 through study completion, an average of 7 months
  Change of days with increased controller (inhaled corticosteroid (ICS) alone or in combination with long-acting bronchodilator (LABA))
Absence days from school/work | Through study completion, an average of 9 months
  Change of absence days from work/school due to asthma
Day-to-day variability of respiratory resistance | Through study completion, an average of 9 months
  Change of average day-to-day coefficient of variation of inspiratory resistance (CVRinsp)
Accuracy of CVRinsp in detecting exacerbations | Through study completion, an average of 9 months
  In the control arm of the study only: accuracy, sensitivity and specificity of day-to-day variability of FOT parameters and of related prediction algorithm in identifying the occurrence of future moderate and severe exacerbations

CONTACTS AND LOCATIONS:
Locations (9):
- Woolcock Institute of Medical Research, Sydney, Australia
- France (2):
  - Grenoble University Hospital, Grenoble
  - University Children's Hospital of Nancy, Nancy
- Italy (6):
  - Azienda Ospedaliero, Universitaria Meyer, Florence, FI
  - AOU Ospedali Riuniti Ancona, Ancona
  - ASST Papa Giovanni XXIII, Bergamo
  - Istituto di Farmacologia Traslazionale (IFT) del CNR, Palermo
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Azienda Unità Sanitaria Locale di Reggio Emilia, Reggio Emilia

IPD SHARING:
Plan to Share IPD: No
No Individual Participant Data (IPD) sharing planned at this stage